CLINICAL TRIAL: NCT07344714
Title: Predicting Respiratory Distress Syndrome in Neonates Delivered in a Lower-Level NICU Setting
Brief Title: Predicting the Need for Prolonged Respiratory Support in Neonates Delivered in a Lower-Level NICU Setting
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William A. Carey, Principal Investigator, Mayo Clinic
Other Study IDs: 24-002867
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome in Premature Infant; Transient Tachypnea of the Newborn; Meconium Aspiration Syndrome; Pneumonia Neonatal; Hyaline Membrane Disease; Pneumothorax; Respiratory Distress Neonatal
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Transient Tachypnea of the Newborn; Meconium Aspiration Syndrome; Hyaline Membrane Disease; Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to analyze the gastric fluid aspirated from the stomachs of neonates receiving routine post-delivery care to predict the need for prolonged respiratory support (>6 hours of life).

DETAILED DESCRIPTION:
The source of the gastric aspirates will be the medical waste generated through the routine care of neonates whose deliveries are attended by the Mayo Clinic neonatal resuscitation team.

ELIGIBILITY:
Inclusion Criteria:

• Both of the following:

* Neonates born at 32 completed weeks gestational age or older whose deliveries are attended by the neonatal resuscitation team and for whom routine gastric suctioning is indicated
* Neonates whose parents actively accepted or did not actively decline the Minnesota Research Authorization.

Exclusion Criteria:

• Any one of the following:

* Neonates with known or suspected congenital anomalies
* Neonates for whom only comfort measures are planned or possible at time of delivery
* Neonates whose parents actively declined the Minnesota Research Authorization.

Ages: 32 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates whose deliveries are attended by the Mayo Clinic neonatal resuscitation team.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance of the algorithmic prediction of the need for prolonged respiratory support, defined as >6 hours of life. | 1 years
  Calculated sensitivity, specificity, positive- and negative-predictive values of the predicted outcomes compared to actual patient outcomes.
Accuracy of algorithmic prediction of negative cases of Respiratory Distress Syndrome | 2 years
  Total proportion of true negatives as determined by the digital point-of-care device algorithm predicting no diagnosis of Respiratory Distress Syndrome and the clinician does not diagnosis Respiratory Distress Syndrome. Reported as a calculation of # true negatives / (# true negatives + # false negatives).

CONTACTS AND LOCATIONS:
Overall Officials: William A. Carey, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leigh BC, Liedl LM, Amsbaugh AL, Carey WA. Spectral analysis of gastric aspirates obtained shortly after birth predicts the need for prolonged respiratory support in neonates in a development cohort. Front Pediatr. 2025 Dec 11;13:1686794. doi: 10.3389/fped.2025.1686794. eCollection 2025. PMID 41458086
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials